CLINICAL TRIAL: NCT03671018
Title: An Open-Label, Randomized, Multicenter, Phase Ib/II Trial Evaluating the Safety, Tolerability, Pharmacokinetics, and Efficacy of Mosunetuzumab (BTCT4465A) in Combination With Polatuzumab Vedotin in Patients With B-Cell Non-Hodgkin Lymphoma
Brief Title: A Study to Evaluate the Safety and Efficacy of Mosunetuzumab (BTCT4465A) in Combination With Polatuzumab Vedotin in B-Cell Non-Hodgkin Lymphoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GO40516; 2018-001141-13 (EudraCT Number)
Record Dates: First submitted 2018-09-10; First posted 2018-09-14 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: B-cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — polatuzumab vedotin; tocilizumab; Rituximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose Finding (Experimental): Participants will receive mosunetuzumab in combination with polatuzumab vedotin. Dose finding will be guided by the observed incidence of dose-limiting toxicities (DLTs) at each dose level.
  Interventions: Drug: Mosunetuzumab (IV); Drug: Polatuzumab vedotin; Drug: Tocilizumab
- Mosunetuzumab + Polatuzumab Vedotin 2L+ R/R FL (Experimental): Participants with at least one line of prior therapy (2L+) and that have relapsed or refractory (R/R) follicular lymphoma (FL) will receive mosunetuzumab + polatuzumab vedotin.
  Interventions: Drug: Mosunetuzumab (IV); Drug: Polatuzumab vedotin; Drug: Tocilizumab
- Mosunetuzumab + Polatuzumab Vedotin 2L+R/R DLBCL (Experimental): 2L+ participants with R/R diffuse large B-cell lymphoma will receive mosunetuzumab + polatuzumab vedotin.
  Interventions: Drug: Mosunetuzumab (IV); Drug: Polatuzumab vedotin; Drug: Tocilizumab; Drug: Rituximab
- Mosunetuzumab SC + Polatuzumab Vedotin 3L+R/R MCL (Experimental): Participants with at least 2 lines of prior therapy (3L+) will receive subcutaneous (SC) mosunetuzumab + polatuzumab vedotin.
  Interventions: Drug: Mosunetuzumab (SC); Drug: Polatuzumab vedotin; Drug: Tocilizumab
- Mosunetuzumab SC + Polatuzumab Vedotin 2L+R/R DLBCL (Experimental): 2L+ participants with R/R DLBCL will receive SC mosunetuzumab and polatuzumab vedotin.
  Interventions: Drug: Mosunetuzumab (SC); Drug: Polatuzumab vedotin; Drug: Tocilizumab

INTERVENTIONS:
Drug: Mosunetuzumab (IV) — Participants will receive intravenous (IV) mosunetuzumab.
  Other Names: BTCT4465A
  Arms: Dose Finding; Mosunetuzumab + Polatuzumab Vedotin 2L+ R/R FL; Mosunetuzumab + Polatuzumab Vedotin 2L+R/R DLBCL
Drug: Mosunetuzumab (SC) — Participants will receive subcutaneous (SC) mosunetuzumab.
  Arms: Mosunetuzumab SC + Polatuzumab Vedotin 2L+R/R DLBCL; Mosunetuzumab SC + Polatuzumab Vedotin 3L+R/R MCL
Drug: Polatuzumab vedotin — Participants will receive IV polatuzumab vedotin.
Drug: Tocilizumab — Participants will receive IV tocilizumab as needed.
Drug: Rituximab — Participants will receive IV rituximab.
  Arms: Mosunetuzumab + Polatuzumab Vedotin 2L+R/R DLBCL

SUMMARY:
This study will evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and efficacy of intravenous (IV) or subcutaneous (SC) mosunetuzumab in combination with polatuzumab vedotin in participants with diffuse large B-cell lymphoma (DLBCL), follicular lymphoma (FL), and mantle cell lymphoma (MCL). It will consist of a dose finding portion followed by an expansion phase for second line or later (2L+) participants with relapsed or refractory (R/R) DLBCL and 2L+ R/R FL. In addition, subcutaneous mosunetuzumab in combination with polatuzumab vedotin will be evaluated in participants with at least 2 prior lines of systemic therapy (3L+) for the treatment of R/R mantle cell lymphoma (MCL) and in participants with 2L+ R/R DLBCL.

ELIGIBILITY:
Key Inclusion Criteria:

* ECOG PS of 0, 1, or 2
* Histologically confirmed FL, DLBCL, or MCL
* Must have received at least one prior systemic treatment regimen containing an anti-CD20-directed therapy for DLBCL or FL
* For MCL, participants must have received at least two prior systemic treatment regiments, which include 1) anti-CD20-directed therapy, 2) BTK inhibitor, and 3) anthracycline or bendamustine
* Relapsed to prior regimen(s) after having a documented history of response (complete response [CR], CR unconfirmed [CRu], or partial response [PR]) of >/= 6 months in duration from completion of regimen(s); or, refractory to any prior regimen, defined as no response to the prior therapy, or progression within 6 months of completion of the last dose of therapy
* Measurable disease, defined as at least one bi-dimensionally measurable nodal lesion, defined as > 1.5 cm in its longest dimension, or at least one bi-dimensionally measurable extranodal lesion, defined as > 1.0 cm in its longest dimension
* Adequate hematologic, renal, and hepatic function

Key Exclusion Criteria:

* Prior treatment with mosunetuzumab or other CD20-directed bispecific antibodies
* Prior treatment with polatuzumab vedotin
* Current > Grade 1 peripheral neuropathy
* Prior use of any monoclonal antibody, radioimmunoconjugate or antibody-drug conjugate (ADC) within 4 weeks before first dose of study treatment
* Treatment with any chemotherapeutic agent, or treatment with any other anti-cancer agent (investigational or otherwise) within 4 weeks or 5 half-lives of the drug, whichever is shorter, prior to first dose of study treatment
* Treatment with radiotherapy within 2 weeks prior to the first dose of study treatment
* Autologous stem-cell transplantation (SCT) within 100 days prior to first study treatment administration
* Prior treatment with chimeric antigen receptor T-cell (CAR-T) therapy within 30 days before first study treatment administration
* Prior allogeneic SCT
* Prior solid organ transplantation
* Known or suspected history of hemophagocytic lymphohistiocytosis (HLH)
* Patients with history of confirmed progressive multifocal leukoencephalopathy (PML)
* Current or past history of central nervous system (CNS) lymphoma or CNS disease
* History of autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 422 (Estimated)
Dates: Start 2018-09-25 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2025-07-20 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Mosunetuzumab in Combination with Polatuzumab Vedotin | Cycle 1 to Cycle 2 (cycle length = 21 days)
Recommended Phase II Dose of Mosunetuzumab in Combination with Polatuzumab Vedotin | Cycle 1 to Cycle 2 (cycle length = 21 days)
Percentage of Participants with Adverse Events (AE) | Baseline through approximately 90 days after last study treatment
Best Objective Response Rate (ORR), Defined as CR or Partial Response (PR) at any Time, Based on PET-CT and/or CT Scan, as Determined by the Independent Review Committee (IRC) using Standard Criteria for NHL | Baseline up to approximately 60 months (assessed at screening and then every 3 months for the first year, then every 6 months until disease progression, start of new anti-cancer therapy, or withdrawal)

SECONDARY OUTCOMES:
Best ORR (CR or PR at any Time) Based on PET-CT and/or CT Scan, as Determined by the Investigator Using Standard Criteria for NHL | Baseline up to approximately 60 months (assessed at screening and then every 3 months for the first year, then every 6 months until disease progression, start of new anti-cancer therapy, or withdrawal)
Best CR Rate on Study Based on PET-CT, and/or CT Scan, as Determined by the Investigator and IRC Using Standard Criteria for NHL | Baseline up to approximately 60 months (assessed at screening and then every 3 months for the first year, then every 6 months until disease progression, start of new anti-cancer therapy, or withdrawal)
CR Rate at the Time of Primary Response Assessment (PRA) Based on PET-CT, as Determined by the Investigator and IRC Using Standard Criteria for NHL | Cycle 8 completion (participants receiving mosunetuzumab), or 5-7 weeks after Cycle 6 (polatuzumab+bendamustine+rituximab participants) (Cycle = 21 days)
ORR, Defined as CR or PR, at PRA Based on PET-CT as Determined by the Investigator and IRC Using Standard Criteria for NHL | Cycle 8 completion (participants receiving mosunetuzumab), or 5-7 weeks after Cycle 6 (polatuzumab+bendamustine+rituximab participants) (Cycle = 21 days)
Duration of Response (DOR) as Determined by the Investigator and IRC Using Standard Criteria for NHL | From the first occurrence of a documented response to disease progression, relapse, or death from any cause, whichever occurs first (up to approximately 60 months)
Progression-Free Survival (PFS) as Determined by the Investigator and IRC Using Standard Criteria for NHL | From time of first study treatment to the first occurrence of disease progression, relapse, or death from any cause, whichever occurs first (up to approximately 60 months)
Event-Free Survival (EFS) as Determined by the Investigator and IRC Using Standard Criteria for NHL | From time of first study treatment to the first occurrence of disease progression, relapse, initiation of new anti-lymphoma treatment (NALT), or death from any cause, whichever occurs first (up to approximately 60 months)
Overall Survival (OS) | From time of first study treatment to death from any cause (up to approximately 60 months)
Anti-Drug Antibodies (ADAs) to Mosunetuzumab | At pre-defined intervals from C1D1 through approximately 90 days after the last study treatment
ADAs to Polatuzumab Vedotin | At pre-defined intervals from C1D1 through approximately 90 days after the last study treatment
Mosunetuzumab Serum Concentration | At pre-defined intervals from C1D1 through approximately 90 days after the last study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (29):
- United States (16):
  - University of Alabama at Birmingham School of Medicine, Birmingham, Alabama
  - City of Hope, Duarte, California
  - University of Colorado Hospital - Anschutz Cancer Pavilion, Aurora, Colorado
  - University of Miami Miller School of Medicine, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - New York University Langone Medical Center, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Lifespan Cancer Institute, Providence, Rhode Island
  - University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Medical College of Wisconsin, Froedtert Hospital;Nephrology Section, Milwaukee, Wisconsin
- Belgium (3):
  - UZ Brussel, Brussels
  - CH Jolimont - Lobbes (Jolimont), Haine-Saint-Paul
  - Clinique St Pierre asbl, Ottignies
- Canada (3):
  - Hamilton Health Sciences - Juravinski Cancer Centre, Hamilton, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - Saskatchewan Cancer Agency (SCA) - Saskatoon Cancer Centre (SCC), Saskatoon, Saskatchewan
- Spain (5):
  - Institut Catala d Oncologia Hospital Duran i Reynals, Barcelona
  - Hospital de San Pedro de Alcantara, Cáceres
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Infanta Leonor; Servicio de Hematologia, Madrid
  - Hospital Universitario Virgen Macarena; Servicio de Oncologia, Seville
- United Kingdom (2):
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Plymouth Hospitals NHS Trust; Pharmacy Dept, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Budde LE, Olszewski AJ, Assouline S, Lossos IS, Diefenbach C, Kamdar M, Ghosh N, Modi D, Sabry W, Naik S, Mehta A, Nakhoda SK, Smith SD, Dorritie K, Jia T, Pham S, Huw LY, Jing J, Wu H, Ead WS, To I, Batlevi CL, Wei MC, Chavez JC. Mosunetuzumab with polatuzumab vedotin in relapsed or refractory aggressive large B cell lymphoma: a phase 1b/2 trial. Nat Med. 2024 Jan;30(1):229-239. doi: 10.1038/s41591-023-02726-5. Epub 2023 Dec 10. PMID 38072960